CLINICAL TRIAL: NCT05137821
Title: Efficacy of Er: YSGG Laser on Oral Biofilm Removal From Implant Surface and Its Biological Response to Periodontal Tissues in Treatment of Peri-implantitis (An Ex Vivo Study)
Brief Title: Efficacy of Er: YSGG Laser in Treatment of Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, alaa, Assistant lecturer of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-REC ID210314
Record Dates: First submitted 2021-10-01; First posted 2021-11-30 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Peri-Implantitis
Keywords: Er: YSGG laser therapy; Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: two group control and test group test group divided into four subgroups
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- non tested comparative group (Experimental): two sealed new implants as a control
  Interventions: Other: no therapy
- Er: YSGG laser tested group (Experimental): 24 infected implants divided into four subgroups that will be decontaminated by Er: YSGG laser in various peri-implant defects
  Interventions: Device: Er: YSGG laser

INTERVENTIONS:
Device: Er: YSGG laser — Er: YSGG laser decontamination of infected implant surfaces to simulate peri-implantitis therapy
  Arms: Er: YSGG laser tested group
Other: no therapy — new sealed implant without any surface treatment
  Arms: non tested comparative group

SUMMARY:
This study will be carried out to evaluate the efficacy of Er: YSGG laser on oral biofilm removal from implant surface in various peri-implant defect morphology in the treatment of peri-implantitis as a primary objective.

To assess the morphological changes and the biological response (biocompatibility) of implant surface after Er: YSGG laser therapy through Profilometer analysis and cell culture process to detect attachment, differentiation, and mineralization of Isolated rat Bone Marrow Mesenchymal stem cells (rBMMSCs) respectively as secondary objectives.

DETAILED DESCRIPTION:
This study will be carried out to evaluate the efficacy of Er: YSGG laser on oral biofilm removal from implant surface in various peri-implant defect morphology in the treatment of peri-implantitis as a primary objective.

To assess the morphological changes and the biological response (biocompatibility) of implant surface after Er: YSGG laser therapy through Profilometer analysis and cell culture process to detect attachment, differentiation, and mineralization of Isolated rat Bone Marrow Mesenchymal stem cells (rBMMSCs) respectively as secondary objectives.

The study was designed as an Ex Vivo study. Four periodontally and systemically healthy volunteers of both gender are included in this study for the formation of in vivo plaque biofilm. Each volunteer will wear a hard resin splint carrying six rough (machined implant; 3.3mm diameter, 8mm length) for 4 days to accumulate dental plaque naturally on the titanium surfaces of the implants.

Therefore, 24 implants will be assessed for Er: YSGG laser therapy in different bone defect simulators.

ELIGIBILITY:
Inclusion Criteria:

* Sex: female or male.
* Age: 25 - 55 years.
* Medically controlled according to medical coding of review of systems (ROS)

Exclusion Criteria:

* Tobacco smoking for at least 6 months before the study enrollment

  * Participants with ill-fitting restorations in both upper first molars that affect the stability of the stent.
  * Participants not following oral hygiene instructions.
  * Participants on dental treatment during the study period.
  * Participants with a history of drug administration
  * Vulnerable group.
  * Participants with long-term mouthwash administration.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
visual inspection of the oral biofilm removal efficacy by image analysis software (Adobe Photoshop | 2 weeks
  evaluate the efficacy of Er: YSGG laser on oral biofilm removal from implant surface in
  various peri-implant defect morphology

SECONDARY OUTCOMES:
Profilometer analysis of surface roughness changes | 1 month
  assess the morphological changes of implant surface after Er: YSGG laser therapy through Profilometer analysis

OTHER OUTCOMES:
biocompatibility test of the surface | 2 months
  assess the biological response (biocompatibility) of implant surface after Er: YSGG laser therapy through cell culture process to detect attachment, differentiation, and mineralization of Isolated rat Bone Marrow Mesenchymal stem cells (rBMMSCs)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Dental School, Cairo, Egypt

REFERENCES:
- [Derived] Hashim A, Kheir El Din NH, El-Khazragy N, Almalahy HG. Comparison of the efficacy of Er,Cr:YSGG laser on oral biofilm removal from implant surfaces with various application times for the treatment of peri-implantitis defects: ex vivo study. BMC Oral Health. 2024 Aug 22;24(1):980. doi: 10.1186/s12903-024-04698-5. PMID 39174958